CLINICAL TRIAL: NCT04973592
Title: Evaluation of Professional Practices in the Management of Blunt Abdominal Trauma in Children in the Pediatric Emergency Department of the Nancy's University Hospital Between 2011 and 2020 : Indentify Children at Low Risk of Intra Abdominal Injuries
Brief Title: Evaluation of Professional Practices in the Management of Blunt Abdominal Trauma in Children in the Pediatric Emergency
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Julie LIENARD, Doctor Julie Lienard - Pediatrician specialized in visceral surgery, Central Hospital, Nancy, France
Other Study IDs: 2020PI292
Record Dates: First submitted 2021-05-12; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Blunt Abdominal Trauma in Children; Identifying Intra Abdominal Injuries
Keywords: Blunt abdominal trauma; Pediatric emergency; Intra-abdominal injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Child with Blunt Abdominal Trauma

SUMMARY:
The aim of our study is primarily to evaluate the professional practices over the last years in the pediatric emergencies of the Nancy's Hospital for the BATiC.

This, in order to identify the traumatic mechanisms and the initial clinical elements which would make it possible to detect the patients at low risk of developing visceral lesions. Then, a management could be proposed which would rationalize the use of additional examinations and would favor the monitoring and the clinical reassessment after the initial management of a minor trauma.

The study of the data will then aim to establish a composite score (anamnestic and clinical) of initial evaluation, from which could result a uniform management protocol (clinical, biological and imaging) of the minor BATiC, of the intermediate BATiC and the major BATiC, applicable to pediatric emergencies at the Nancy's Hospital.

DETAILED DESCRIPTION:
For children aged 1 to 18, trauma is one of the leading causes of death, ahead of cancer and congenital malformations. The traumatic mechanisms are mainly accidents on public roads (car accidents, two-wheel accidents, accidents involving a pedestrian), sports accidents (especially cycling and horse riding), falls from a high height or onto a blunt object, and intentional or unintentional direct hits. Mortality is mainly correlated with involvement of the skull, thorax and abdomen and there is a clear male predominance (sex ratio 2 to 3 boys / 1 girl).

In France, blunt abdominal trauma in children (BATiC) is a frequent reason for consultation in pediatric emergencies. It accounts for 20 to 30% of childhood trauma, among which 10 to 30% result in potentially life-threatening intra-abdominal injuries (IAI). In order of frequency, the organs most affected are the spleen, the liver, kidneys and the pancreas. Rarely, hollow organs such as the small intestine, the duodenum, the colon, or the stomach can be affected. In rarer occasion, sores of the mesentery may be seen to.

BATiC is opposed to penetrating abdominal trauma, which accounts for only 5 to 15% of abdominal trauma in children. It is frequently part of a multiple trauma defined by "a child who has suffered a trauma whose kinetics are likely to cause at least two lesions, at least one of which can be life-threatening".

While multiple trauma accounts for only 14% of childhood trauma, it is nonetheless the main cause of death after the age of 1. For several years, this has motivated the establishment of emergency treatment protocols under the impetus of the development of "trauma centers". Therefore, polytrauma has well-codified diagnostic criteria and precise and systematic management, applicable to pediatric emergencies. Regarding the isolated BATiC, the management is less unequivocal. Although it is more frequent, BATiC with low or medium kinetics does not benefit from any clear management protocol.

Indeed, the management of a child admitted for BATiC in the pediatric emergency room does not necessarily take into account the traumatic mechanism. The course of action currently adopted involves at least an initial clinical evaluation, sometimes repeated after a period of monitoring. Then it is frequently supplemented by the performance of a blood test and imaging aimed at detecting possible IAI.

In current practice, some practitioners choose this systematic approach of BATiC, including complementary examinations from the outset, in order to never ignore an IAI. Others seem to support a more reserved attitude to the use of complementary exams when the initial assessment is reassuring. It is clear that many abdominal traumas are not complicated by any visceral injury. Especially when the traumatic mechanism is minimal and when the initial clinical evaluation does not identify elements of seriousness. In these different situations, carrying out additional examinations may indeed seem excessive.

Therefore, there is a great heterogeneity of BATiC and a strongly practitioner-dependent care which does not always take into account the minor traumatic mechanism.

Establishing a validated management protocol for BATiC, as can be the case with polytrauma, is difficult due to the great diversity of traumatic mechanisms and their variable kinetics. All the more so since the same mechanism does not systematically expose people to the same lesions depending on the child's age and its morphological characteristics. It is fundamental to take into consideration the anatomical and physiological specificities of the growing child which define his fragility in the face of abdominal trauma. Another difficulty lies in the anamnestic collection of facts which may be limited due to the child's age, his apprehension (hospital environment, reaction of the caregiver), the medical context (general condition, underlying pathology, psychological state) and the social context (particular case of mistreatment). This is all the more difficult when the trauma is not seen by a third party at all.

Several studies have already sought to define predictive scores for IAI. These scores are established after performing additional laboratory tests and almost always include performing an abdominal ultrasound. They have the advantage of reducing the use of the scanner, thus exposure to ionizing rays, but do not simplify the management of minor trauma for which it would be possible not to perform additional examinations at all, if they are defined beforehand.

Retrospective study of the anamnestic and clinical elements of patients without any IAI could allow the identification of clinical situations in which the performance of complementary examinations is not necessary. In this way, the course of action for minor trauma could be simplified by promoting surveillance and clinical reassessment rather than the routine use of additional tests, thereby reducing the time spent in the pediatric emergency room.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 0 to 18 years consulting the Pediatric Emergency Department of the Nancy University Hospital.
* Primary care
* Blunt abdominal trauma

Exclusion Criteria:

* Secondary management
* Polytrauma
* Open abdominal trauma / Penetrating wound
* Polyhandicap
* Pre-existing major digestive or urinary pathology (single kidney, renal or hepatic transplantation...)
* Pre-existing hemostasis or hepatic disorders or trauma (inborn or acquired causes)

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients under 18 years of age who consulted the pediatric emergency department of the Nancy University Hospital between 08/03/2011 (first date of use of resurgences) and 22/09/2020 (end date of collection for the study) for closed abdominal trauma.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Characteristics of the blunt abdominal trauma studied : Trauma mechanisms | Day 0
  fall from a bicycle, a horse, a height, road - belted or unbelted accident, two-wheeler accident, blows inflicted
Characteristics of the blunt abdominal trauma studied : Trauma kinetics | Day 0
  low (< 50km/h) or high (> 50km/h)
Clinical evaluation : Pain | Day 0
  visual analog scale : 0 to 10
Clinical evaluation : Location of pain | Day 0
  9 abdominal quadrants
Clinical evaluation : Type of pain | Day 0
  pain, defense or contracture
Hemodynamic evaluation : Heart rate | Day 0
  beat/min
Hemodynamic evaluation : Blood pressure | Day 0
  mmHg
Hemodynamic evaluation : Respiratory rate | Day 0
  cycle/min

SECONDARY OUTCOMES:
Demographic criteria of the study population : Age | Day 0
  in months
Demographic criteria of the study population : Gender | Day 0
  male or female
Time to management : Time between trauma and consultation | Day 0
  minutes Management time (medical evaluation, blood work, imaging)
Time to management : Management time | Day 0
  medical evaluation, blood work, imaging
Biological examinations : Blood count | Day 0
  g/dL
Biological examinations : Liver enzyme | Day 0
  UI/L
Biological examinations : Pancreatic enzyme | Day 0
  UI/L
Biological examinations : Coagulation test | Day 0
  prothrombin time
Biological examinations : Blood group | Day 0
  G/L
Imaging examinations : Imaging | Day 0
  body scanner, abdominal-pelvic scanner or ultrasound
Imaging examinations : Imaging findings | Day 0
  presence of an effusion, hollow organ or solid organ lesion + AAST classifications
Surgical advice | Day 0
  Surgical opinion required
Orientation | Day 0
  Return home or Hospitalization Hospitalization (surgery,intensive care)
Type of management | Day 0
  Medical or surgical management
Second consultation at emergency | 30 days
  Consultation (within 1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Marine Pettini, Principal Investigator
Locations (1):
- Marine Pettini, Nancy, France